CLINICAL TRIAL: NCT01330199
Title: A Phase I Investigation of Single-Dose Pharmacokinetics of Tenofovir, Emtricitabine, Maraviroc, and Raltegravir in Cervical, Vaginal, and Rectal Tissues and Secretions
Brief Title: Pharmacokinetics of Tenofovir, Emtricitabine, Maraviroc, and Raltegravir in Cervical, Vaginal, and Rectal Tissues and Secretions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Responsible Party: Principal Investigator, Angela Kashuba, PharmD, Professor, University of North Carolina, Chapel Hill
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 10-1393
Record Dates: First submitted 2010-08-17; First posted 2011-04-06 (Estimated); Last update posted 2013-09-17 (Estimated); Status verified 2013-09

CONDITIONS: Healthy Adult Females
Keywords: Healthy; Female; Volunteer

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- TDF 150mg + MVC 150mg (Experimental): Subjects will receive a single dose of tenofovir 150 mg and maraviroc 150 mg.
  Interventions: Other: Pharmacokinetic Sampling
- TDF 300mg + MVC 300mg (Experimental): Subjects will receive a single dose of tenofovir 300 mg and maraviroc 300 mg.
  Interventions: Other: Pharmacokinetic Sampling
- TDF 600mg +MVC 600mg (Experimental): Subjects will receive a single dose of tenofovir 600 mg and maraviroc 600 mg.
  Interventions: Other: Pharmacokinetic Sampling
- FTC 100mg + RAL 200mg (Experimental): Subjects will receive a single dose of emtricitabine 100 mg and raltegravir 200 mg.
  Interventions: Other: Pharmacokinetic Sampling
- FTC 200mg + RAL 400mg (Experimental): Subjects will receive a single dose of emtricitabine 200 mg and raltegravir 400 mg.
  Interventions: Other: Pharmacokinetic Sampling
- FTC 400mg + RAL 800mg (Experimental): Subjects will receive a single dose of emtricitabine 400 mg and raltegravir 800 mg.
  Interventions: Other: Pharmacokinetic Sampling

INTERVENTIONS:
Other: Pharmacokinetic Sampling — Blood plasma, Rectal, Cervical, and Vaginal Tissues and Secretions

SUMMARY:
The purpose of this study is to develop a predictive antiretroviral pharmacokinetic model of mucosal fluid and tissue distribution in genital tract fluid, rectal fluid and 3 mucosal tissues. This will be accomplished by determining the pharmacokinetic disposition and dose proportionality of four antiretrovirals (tenofovir, emtricitabine, maraviroc, and raltegravir) in human rectal and cervicovaginal fluid and rectal, cervical, and vaginal tissue.

ELIGIBILITY:
Inclusion Criteria:

* Healthy pre-menopausal female subjects between the ages of 18 and 49 years, inclusive, with an intact gastrointestinal tract, uterus, and cervix. (Healthy is defined as no irregular menstrual cycles or clinically relevant abnormalities identified by a detailed medical history, full physical examination, including blood pressure and pulse rate measurement, 12-lead ECG and clinical laboratory tests.)
* All subjects must have an estimated calculated creatinine clearance of at least 80 mL/min by the Cockcroft-Gault formula
* All subjects must have a negative serum pregnancy test at screening and negative urine pregnancy tests on days of sampling and should be using at least one of the following methods of contraception:
* Systemic hormonal contraceptive (oral, depot, transdermal or implant)
* IUD placed at least 1 month prior to study enrollment
* Bilateral tubal ligation (Sterilization)
* Vasectomized male partner
* Condom + Spermicide

  *Unless engaged in sexual activity with female only sex partners or abstinent for at least 3 months prior with no intention of becoming sexually active during the study period. Any history of recent or present concomitant male sex partners will be addressed and ruled out in the context of screening participants for eligibility for the protocol
* Female only partner
* Body Mass Index (BMI) of approximately 18 to 34 kg/m^2; and a total body weight > 45 kg (99 lbs).
* Evidence of a personally signed and dated informed consent document indicating that the subject has been informed of all pertinent aspects of the trial.
* Willing and able to comply with scheduled visits, treatment plan, laboratory tests, and other trial procedures.
* Subject must have a normal pap smear within 36 months of the screening visit, no procedures for abnormal cervical/vaginal pathology in the last six months, at least one prior gynecological visit as part of subject's routine medical history.
* Subject must be willing to abstain from sexual intercourse, douching, and all intravaginal and intrarectal products at least 72 hours prior to Day 1 until study completion.
* Subject must be HIV-1 and Hepatitis B surface antigen negative as documented on screening labs.
* Subject must not be actively involved in the conception process.
* Subject must be able to swallow pills and have no allergies to any component of the study products.

Exclusion Criteria:

* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic, or allergic disease (including documented drug allergies, but excluding untreated, asymptomatic, seasonal allergies at time of dosing).
* Subjects with a history of hysterectomy
* Subjects who are pregnant, possibly pregnant, or lactating
* Subjects with a presence of vaginal discharge or genital bleeding at screening
* History of febrile illness within five days prior to first dose.
* Any condition possibly affecting drug absorption (eg, gastrectomy).
* A positive urine drug screen.
* A positive result for HIV.
* Active Hepatitis B infection as determined by positive Hepatitis B surface antigen (HbsAg) or Hepatitis B core antibody (HBcAb) tests (in the absence of HBsAb).
* Active Hepatitis C infection as defined by anti-hepatitis C virus serology (determined by multi-antigen EIA) and detectable Hepatitis C viral RNA.
* A positive test for syphilis, gonorrhea, Chlamydia, or trichomonas at screening or symptomatic bacterial vaginosis.
* Any laboratory chemistry or hematology result Grade 2 or greater according to the DAIDS Laboratory Grading Tables.
* Treatment with an investigational drug within 4 months preceding the first dose of trial medication.
* History of regular alcohol consumption exceeding 14 drinks (1 drink = 5 ounces (150 mL) of wine or 12 ounces (360 mL) of beer or 1.5 ounces (45 mL) of spirits) per week.
* Participation in a clinical trial involving vaginal or rectal biopsies within 12 months preceding the first dose of trial medication.
* Use of prescription or nonprescription drugs, vitamins, and dietary supplements within 7 days or 5 half-lives (whichever is longer) prior to the first dose of trial medication. As an exception, systemic hormonal methods of contraception can be continued.
* Blood donation of approximately 1 pint (500 mL) within 56 days prior to dosing
* History of sensitivity to heparin or heparin-induced thrombocytopenia
* Any vaccination within 30 days of study entry
* Allergy to lidocaine or Mohl's solution
* Allergy to latex
* Abnormal pap smear in the past 12 months
* Any degree of ectopy or abnormality evident during the pelvic exam at screening
* Any condition which, in the opinion of the investigator, is likely to interfere with follow-up or ability to take the study medication appropriately.
* Unwilling or unable to comply with the following dietary restriction in regard to study drug administration:
* Subjects must abstain from all food and drink (except water) at least 4 hours prior to any safety laboratory evaluations
* Subjects must abstain from all food and drink (except water) at last 8 hours prior to the start of pharmacokinetic sample collections
* Subjects will not be allowed to eat or drink grapefruit containing products from 7 days prior to the first dose of trial medication until collection of the final pharmacokinetic blood sample. While confined, the total daily nutritional composition will be approximately 50% carbohydrate, 35% fat and 15% protein, and the daily caloric intake per subject should not exceed approximately 3200 kcal.
* Subjects will be required to consume only a clear liquids diet the night before the rectal biopsy procedure and until the procedure has been completed

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 49 (Actual)
Dates: Start 2012-02; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Dose Proportionality | 48 hours
  To determine if antiretroviral mucosal fluid and tissue concentrations change proportionally with a change in antiretroviral dose.

CONTACTS AND LOCATIONS:
Overall Officials: Angela DM Kashuba, PharmD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- UNC Hospitals CTRC, Chapel Hill, North Carolina, United States